CLINICAL TRIAL: NCT01320228
Title: Effect of Dietary Components on Gastrointestinal Side Effects Induced by Orlistat, a Lipase Inhibitor
Acronym: ORLIFAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Arne Astrup, Professer, Dr. Med., University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: B274
Record Dates: First submitted 2011-03-21; First posted 2011-03-22 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Obesity
Keywords: Obesity; orlistat; fat excretion; fiber; dairy calcium
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Placebo Comparator): Alli treatment plus placebo (rice flour)
  Interventions: Dietary Supplement: Control
- Capolac (Experimental): Alli treatment plus Capolac supplement (1200 Ca/d from Capolac)
  Interventions: Dietary Supplement: Capolac
- Flax fiber (Experimental): Alli treatment plus flaxseed fibers (5 g/d of dietary fibers from flaxseed)
  Interventions: Dietary Supplement: Flax fiber
- Capolac+Flax fiber (Experimental): Allit treatment plus Capolac (1200 mg Ca/d from Capolac) and Flax fiber (5 g dietary fiber from flaxseed)
  Interventions: Dietary Supplement: Capolac+Flax fiber

INTERVENTIONS:
Dietary Supplement: Control — Alli treatment plus placebo (rice flour)
  Arms: Control
Dietary Supplement: Capolac — Alli treatment plus Capolac supplement (1200 Ca/d from Capolac)
  Arms: Capolac
Dietary Supplement: Flax fiber — Alli treatment plus flaxseed fibers (5 g/d of dietary fibers from flaxseed)
  Arms: Flax fiber
Dietary Supplement: Capolac+Flax fiber — Allit treatment plus Capolac (1200 mg Ca/d from Capolac) and Flax fiber (5 g dietary fiber from flaxseed)
  Arms: Capolac+Flax fiber

SUMMARY:
The objective of the Orlifat trial is to investigate if dietary fibres from linseeds and dairy calcium (Capolac ®) may reduce gastrointestinal side effects related to increased fecal fat content, induced by treatment with Alli® (orlistat). Secondly, effect on food intake, anthropometry, Quality of Life and cardiovascular risk markers will be evaluated. The trial is designed as a randomised 2 x 2 factorial 13-weeks parallel intervention, in which 72 obese participants will be randomised to supplementation with flaxseed fibres and/or dairy calcium concentrate (Capolac) in addition to treatment with Alli ®:

1. Alli® (60 mg t.i.d) plus placebo (rice flour)
2. Alli® plus 5 g flaxseed fibers
3. Alli® plus 1200 mg Ca from Capolac
4. Alli® plus 5 g flaxseed fibers and 1200 mg Ca from Capolac

ELIGIBILITY:
Inclusion Criteria:

* 20-60 years of age
* men and women
* BMI 30-40 kg/m2

Exclusion Criteria:

* Dairy allergy and/or intolerance, allergy to Orlistat
* Infectious and metabolic diseases
* Gastrointestinal diseases (previous and current)
* Troubles swallowing tablets and capsules
* Dietary supplement use during the trial and 1 month prior to the trial
* Postmenopausal (selfreported)
* Pregnancy and lactation
* Treatment with oral anticoagulation medications, ciclosporin, levothyroxin, antiepileptika, acarbose and amiodaron
* Prescription medication will be considered on an individual basis at the screening visit according to SOP
* Dieting or other changes of diet within 3 months
* Participation in other trials

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Ratings of gastrointestinal comfort | baseline, week 0, 2, 4, 8, 12
  Subjective assessment of gastrointestinal comfort using visual analogue scales

SECONDARY OUTCOMES:
Total fecal fat excretion | week 0 and 4
  Average total fecal fat excreted during five days in week 0 and week 4
Total, LDL and HDL cholesterol | baseline and 12
Ratings of quality of life | baseline, week 0, 2, 4, 8 and 12
  Questionnaire used to assess quality of life related to obesity and treatment thereof
Body weight | baseline, week 0, 2, 4, 6, 8, 10 and 12
Waist and hip circumference | Baseline, week 0, 2, 4, 6, 8, 10 and 12
food intake | week 0 and 4
  Intake of total fat and energi estimated using 7d weighed food records
Habitual intake of dietary fiber and calcium | baseline
  Habitual intake of dietary fiber and calcium estimated using food frequency questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, MD, Dr.med., Study Director — Department of Human Nutrition, Faculty of Life Sciences, University of Copenhagen
Locations (1):
- Department of Human Nutrition, Faculty of Life Sciences, University of Copenhagen, Frederiksberg C, Denmark

REFERENCES:
- [Derived] Kristensen M, Juul SR, Sorensen KV, Lorenzen JK, Astrup A. Supplementation with dairy calcium and/or flaxseed fibers in conjunction with orlistat augments fecal fat excretion without altering ratings of gastrointestinal comfort. Nutr Metab (Lond). 2017 Feb 7;14:13. doi: 10.1186/s12986-017-0164-8. eCollection 2017. PMID 28191026